CLINICAL TRIAL: NCT04276350
Title: Efficacy of Acupuncture as a Treatment for Faecal Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Singapore College of Traditional Chinese Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/2525
Record Dates: First submitted 2020-02-18; First posted 2020-02-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Faecal Incontinence
Keywords: Acupuncture; Faecal Incontinence; Traditional Chinese Medicine
MeSH Terms: conditions — Encopresis | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture Regime:
  2-3 sessions per week, each lasting an hour, over a period of 10 weeks (with deviation of 2 weeks for scheduling), total of 30 sessions
  Interventions: Procedure: Acupuncture
- Best medical therapy (Active Comparator): Best Medical Therapy Regime:
  3 sessions to be completed over a period of 10 weeks (with deviation of 2 weeks for scheduling), with subjects learning and practicing biofeedback exercises daily
  Interventions: Procedure: Best Medical Therapy

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture sessions - 2-3 times/week, each session lasting 1 hour, over a period of 10 weeks (with allowed deviation up to 2 weeks due to scheduling)
  Arms: Acupuncture
Procedure: Best Medical Therapy — Best Medical Therapy - 3 biofeedback sessions over a period of 10 weeks (with allowed deviation up to 2 weeks due to scheduling), where subjects learn and practice the exercises daily
  Arms: Best medical therapy

SUMMARY:
Overall Aim:

To improve the long-term management outcomes for faecal incontinence (FI); through the implementation of new alternative treatment to complement existing treatment options, and enable better utilization of limited healthcare resources.

Primary Specific Aim:

To evaluate the effectiveness of Traditional Chinese Medicine (TCM) acupuncture in the treatment of faecal incontinence.

Secondary Aims:

* To evaluate the safety profile of TCM acupuncture.
* To explore the patient satisfaction and uptake of TCM acupuncture as an alternative management strategy for FI.
* To evaluate improvements in health-related quality of life with TCM-acupuncture.
* To explore the cost-effectiveness of TCM acupuncture.

Hypothesis:

Traditional Chinese Medicine therapy, in the form of acupuncture, is an effective treatment for faecal incontinence.

DETAILED DESCRIPTION:
Experimental design and procedure The study will run as a prospective, multi-centre, randomised controlled trial of patients with faecal incontinence of best medical therapy versus TCM-Acupuncture.

Patient reported outcome measures and assessments will be carried out to assess primary and secondary outcomes at the commencement of trial, after 10 weeks of the intervention, then again at 15 weeks.

Recruitment procedure Patients will be recruited from Singapore General Hospitals' Colorectal Surgery Department. SGH possess a fully staffed pelvic floor unit specialising in the treatment of faecal incontinence. Eligible patients will be assessed and counselled by a member of the colorectal surgical team. They will then attend for consenting and baseline assessment.

The clinicians will inform the patient during the initial consultation about the different treatments available for their condition as well as this study. As is normal clinical practice, the clinicians will explain the risks and benefits of all the treatment options. Each potential participant will be provided with a patient information sheet. Those who consent to inclusion will then be contacted by a member of the research team. Informed consent will be taken in the clinic environment.

Randomisation Patients will be randomised into one of two groups, to receive acupuncture treatment (INTERVENTION GROUP) or to have best medical therapy (BMT) (CONTROL GROUP). Both patients in the INTERVENTION GROUP and CONTROL GROUP will continue their previous medication, if any, throughout the duration of the study. This is to standardise the 'steady-state' existing in this often elderly population, already subject to polypharmacy.

Patients in the INTERVENTION GROUP will undergo acupuncture therapy at the Singapore College of Traditional Chinese Medicine (SC-TCM), performed by a team of TCM practitioners regularly using acupuncture in the treatment of faecal incontinence and bowel conditions. This regimen will comprise 3 sessions per week each lasting 1 hour, over a period of 10 weeks, for a total of 30 sessions.

Patients in the CONTROL GROUP will undergo BMT as defined previously for the same period of 10 weeks.

Patients will be asked to maintain a simple bowel diary, and answer the FIQL and St Marks' incontinence scores at weeks 0, 10, and 15 to record the primary and secondary outcome measurements. Anorectal Physiology will be offered to patients at 0 and 10 weeks, but for the purposes of this study protocol, will be purely voluntary. We understand that this invasive examination would be a significant undertaking and potential barrier to recruitment for many patients.

Follow up procedure Patient follow-up will consist of three visits to the hospital following the randomisation to either arm of the study. This will be at the 5 week period, 10 week period and 15 week period of the study, where the primary and secondary outcomes measurements will be assessed.

Randomisation and allocation Participants will be randomised to one of the two study groups in equal proportion using a blinded bag shuffling method. This will take place upon agreement to participate.

Measures of outcome Primary outcome: Bowel diary - Incontinence episodes per week Secondary outcomes: St Marks' incontinence score, Faecal Incontinence Quality of Life (FIQL) score, Anorectal manometry scores (at week 0, and 10 weeks) - optional for participants. Analysis plans and sample size sought The primary end-point of the study was defined as the difference in weekly faecal incontinence episodes when comparing patients randomized to the INTERVENTION and CONTROL arms. The secondary endpoint of the study was defined as the difference in St Marks' score and FIQL when comparing patients randomized to the INTERVENTION and CONTROL arms.

Sample Size To detect a difference of 30% between the two arms, assuming that the proportion of incontinence episodes in the conservative arm is 20%, a total sample size of 90 will be required at alpha=0.05 with 80% power. Accounting for a drop-out rate of 10%, the total sample size required is 100, to be recruited over 30 months.

Statistical analysis Continuous data will be summarized as mean (SD) or median (IQR) as appropriate and categorical/binary data as frequency (%). Statistical significance will be set at 0.05. Intention to treat (ITT) analysis will be performed.

The primary hypothesis will be evaluated using a Chi-square test or a Fisher's exact test as appropriate. Additionally, we will also model the outcome using a generalized linear model with a logit link. The possible treatment effect modification of clinically important factors (age, gender, ASA status) will be evaluated in the model.

The secondary hypothesis to evaluate the St Marks' score will be assessed using a two-sample t-test assuming that the score can be treated as a continuous measure. The difference in the FIQL between the two arms will also be tested using the two-sample t-test.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with faecal incontinence
* At least 2 episodes of faecal incontinence per week, St Mark's incontinence score of 5 or greater
* Patients aged 21 years or older
* Prior colonoscopy done to exclude underlying colonic pathology
* Written informed consent obtained

Exclusion Criteria:

* Active inflammation of the bowel, including inflammatory bowel disease, infection or perianal sepsis
* Pregnant women
* Current or previous diagnosis of the gastrointestinal tract, genitourinary, or pelvic cancers
* Presence of congenital or acquired neurological deficits (including spinal disorders)
* Previous history of complex major pelvic, anal or rectal surgery
* Previous history of multi-focal or major sphincter injuries or deficits

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who showed improvement in weekly number of incontinence episodes (baseline compare to subjects' week 10) | 10 weeks
  Assessed for superiority of intervention arm compared to the control arm

SECONDARY OUTCOMES:
Mean change in St Mark's incontinence score | 10 weeks
  Mean change in St Mark's incontinence score at week 10 from baseline (superiority comparison)
Mean change in Faecal Incontinence Quality of Life (FIQL) score | 10 weeks
  Mean change in Faecal Incontinence Quality of Life (FIQL) score at week 10 from baseline (superiority comparison)

OTHER OUTCOMES:
Mean change in anorectal manometry scores | 10 weeks
  Mean change in anorectal manometry scores at week 10 from baseline (superiority comparison)

CONTACTS AND LOCATIONS:
Overall Officials: Emile Kwong Wei Tan, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Ng YY, Tan KY, Zhao Y, Seow-En I, Chok AY, Chuang J, Loy MS, Tan EK. Efficacy of Traditional Acupuncture Compared to Biofeedback Therapy in Fecal Incontinence: A Randomized Controlled Trial. Dis Colon Rectum. 2024 Oct 1;67(10):1313-1321. doi: 10.1097/DCR.0000000000003357. Epub 2024 Jul 2. PMID 38954475